CLINICAL TRIAL: NCT02534103
Title: Relationship Between a Combined Index of Diastolic and Systolic Performance and Intraoperative Hemodynamic Changes During Off-pump Coronary Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0879
Record Dates: First submitted 2015-07-23; First posted 2015-08-27 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Obstructive Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
As considering the close relationship between systolic dysfunction and diastolic dysfunction, the EAS index e'/(a' x s') including systolic and diastolic function could be expected to predict hemodynamic changes during off-pump coronary artery bypass surgery(OPCAB). Exposure of the grafting site during OPCAB needs displacement of the heart, resulting in hemodynamic instability.

Therefore the investigators are going to evaluate EAS index with preoperative Transthoracic echocardiography(TTE) and want to know the relationship between preoperative EAS index and intraoperative hemodynamic changes in patients undergoing OPCAB, in a prospective observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20
2. Patients undergoing multivessel off-pump coronary artery bypass surgery

Exclusion Criteria:

1. Age < 20
2. Patients with valvular heart disease
3. Congestive heart failure, NYHA class ≥III
4. Emergency surgery
5. Patients with arrhythmia
6. ST segment elevation myocardial infarction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery obstructive disease planned to have multivessel OPCAB
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-08-04; Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
sequential changes of SvO2 | during OPCAB surgery
  Mixed venous oxygen saturation(SvO2) reflects the balance of oxygen supply and demand immediately. Cardiac index(CI) also is a useful marker of how well the heart is functioning. Both variables can show the hemodynamic instability. With the comparison of EAS index and variables including SvO2 and CI, Investigator may draw the predictable value of the EAS index for predicting hemodynamic instability during OPCAB.
sequential changes of CI | during OPCAB surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kwang Shim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea